CLINICAL TRIAL: NCT04926428
Title: In Situ Thrombolysis With tPA and Inflow Lung Perfusion Analysis in Patient With Severe Covid-19 Infection
Brief Title: In Situ Thrombolysis With tPA and Inflow Perfusion Analysis in Patient With Severe Covid-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Mexicano para el Estudio de la Medicina Intensiva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DI-222-2020
Record Dates: First submitted 2021-06-13; First posted 2021-06-15 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: Covid-19; Acute Respiratory Distress Syndrome; Thrombosis
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): In situ thrombolysis with tPA
  Interventions: Drug: tPA

INTERVENTIONS:
Drug: tPA — Selectively catheter thrombolysis with alteplase in each main pulmonary
  Other Names: in situ thrombolysis

SUMMARY:
To estimate the pulmonary response microvascular thrombosis in critical patients due to SARS-Cov-2., at the Hospital General de México "Dr. Eduardo Liceaga", a 15 patients compassionate treatment study was authorized and approved by the ethics and research committee DI-222-2020. Because of the severity of the illness the legal representative sign informed consent in all the patients for performing in-situ thrombolysis with alteplase selectively by catheter in each main pulmonary artery, under fluoroscopic guidance and acquiring images with the iFlow software to assess immediate and post-procedure response.

DETAILED DESCRIPTION:
The main clinical characteristic of patients with severe SARS-Cov-2 infection is hypoxemic respiratory failure that requires Mechanical Ventilation. The Acute Respiratory Syndrome model has been proposed as the cause of this significant deterioration in lung function and all management has focused on ventilatory support management. As for ventilatory failure, it has been attributed to the presence of severe pulmonary inflammation evolving to fibrosis, which is the clinical characteristic of patients with Primary Respiratory Distress Syndrome (which would be the case of this as it is considered a respiratory virus).

Several autopsy studies demonstrated microthrombi in pulmonary circulation. The major limitation of these investigations is that the autopsy provided static information. Some of these alterations could be secondary to the disseminated intravascular coagulation (DIC) observed as the standard route to the multisystem organ failure exhibited in critically ill patients.

With this comes the contradictory results of high doses of anticoagulants in the survival of these patients. This intermediate to high doses can reduce organ support treatments in moderate cases, however, in critically ill patients the benefit of high dose of anticoagulants, once again failed to produce benefit on survival. Different publication on biopsies made in these patients have report the presence of thrombosis in the microcirculation and finally recently has been published the demonstration by direct examination with Citoscam, the presence of this thrombosis of the microcirculation in vivo in 11 of 13 test (85% of the sample). Studies performed with viscoelastic coagulation tests present evidence of three key alterations in coagulation

1. EXTEM and INTEM Hypercoagulable states represented by a maximum amplitude (A5, A10 and MCF) greater than 70mm, short clot formation time.
2. Hyperfibrinogenemia A5 A10 MCF in FIBTEM greater than 30mm
3. Absence of fibrinolytic activity (ML% Lys 30 and Lys 60) 100% Taking this into account plus the large number of publications regarding the thrombotic phenomenon of the patient with COVID-19, this could be explained by the presence of a phenomenon of ventilation perfusion (V / Q) that is observed in patients with Massive Pulmonary Thromboembolism (PE) which is known as the infinite relationship, that is, the lung is with normal aeration, but no perfusion, there is no adequate gas exchange, with presence of hypoxia, increment of death space and ultimately obstructive shock.

In patients with COVID-19, this phenomenon is observed in patients with absence of massive or submassive PE that explains this phenomenon.

The high mortality of critically ill patients with SARS-Cov-2 infection, the presence of thrombosis of the microcirculation and the lack of efficacy of anticoagulation in some cases suggests that this phenomenon could be the cause of the behavior between perfusion ventilation observed in SARS-Cov-2 patients.

For these reasons, a probe of concept research was developed to find out if pulmonary perfusion alteration by microthrombosis and secondary V / Q abnormalities could be linked to the pathophysiology of the patient with severe SARS-Cov-2 infection.

To estimate the pulmonary response microvascular thrombosis in critical patients due to SARS-Cov-2., at the Hospital General de México "Dr. Eduardo Liceaga", a 15 patients compassionate treatment study was authorized and approved by the ethics and research committee DI-222-2020. Because of the severity of the illness the legal representative sign informed consent in all the patients for performing in-situ thrombolysis with alteplase selectively by catheter in each main pulmonary artery, under fluoroscopic guidance and acquiring images with the iFlow software to assess immediate and post-procedure response.

ELIGIBILITY:
Inclusion Criteria:Lung criteria:

Patients with severe Covid 19 nfection, from 18 to 75 years old, Invasive Mechanical Ventilation (IMV) Pao2 / fio2 less than 150 Non réponse to prone position Coagulation criteria ISTH score >5, D-dimer greater than 1200, Viscoelastic testing EXTEM A5 >65 FIBTEM > 30 and EXTEM ML<8%

-

Exclusion Criteria:

Ischemic CVD or presence of abnormal neurological examination. Active bleeding. Acute Myocardial Infarction within the previous three weeks or cardiac arrest during hospitalization.

cardiac tamponade. endocarditis. uncontrolled hypertension SBP> 185mmhg or DBP> 110. history of stage 4 cancer. history of brain tumor. Arterious venous malformation ruptured aneurysm. major surgery in the previous 2 weeks major trauma in the previous 2 weeks. pregnancy. fibrinogen less than 200 blood dyscrasias thrombocytopenia less than 30,000

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in lung perfusion | 1 hour
  changes in contrast distribution comparing pre and post-thrombolysis using Iflow parameters that include ROI, peak flow and Time

SECONDARY OUTCOMES:
Coagulation | 48 hours
  changes in D Dimer, standard coagulation test and fibrinogen
Oxygenation Index | 48 hours
  changes in PaO2/FiO2 index pre and post-thrombolysis

CONTACTS AND LOCATIONS:
Overall Officials: Jose Damian Carrillo Ruiz, PhD, Study Director — Hospital General de Mexico Dr. Eduardo Liceaga
Locations (1):
- Hospital General de Mexico Dr Eduardo Liceaga, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared by petition.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months up to 5 years after completion
Access Criteria: proposal should be directed to gmemiinv@gmails.com, to gain access, requestor will need to sign a data access agreement

REFERENCES:
- [Background] Greene R. Pulmonary vascular obstruction in the adult respiratory distress syndrome. J Thorac Imaging. 1986 Jul;1(3):31-8. doi: 10.1097/00005382-198607000-00006. PMID 3298679
- [Background] Yao XH, Li TY, He ZC, Ping YF, Liu HW, Yu SC, Mou HM, Wang LH, Zhang HR, Fu WJ, Luo T, Liu F, Guo QN, Chen C, Xiao HL, Guo HT, Lin S, Xiang DF, Shi Y, Pan GQ, Li QR, Huang X, Cui Y, Liu XZ, Tang W, Pan PF, Huang XQ, Ding YQ, Bian XW. [A pathological report of three COVID-19 cases by minimal invasive autopsies]. Zhonghua Bing Li Xue Za Zhi. 2020 May 8;49(5):411-417. doi: 10.3760/cma.j.cn112151-20200312-00193. Chinese. PMID 32172546
- [Background] Livingston E, Bucher K. Coronavirus Disease 2019 (COVID-19) in Italy. JAMA. 2020 Apr 14;323(14):1335. doi: 10.1001/jama.2020.4344. No abstract available. PMID 32181795
- [Background] Vesconi S, Rossi GP, Pesenti A, Fumagalli R, Gattinoni L. Pulmonary microthrombosis in severe adult respiratory distress syndrome. Crit Care Med. 1988 Feb;16(2):111-3. doi: 10.1097/00003246-198802000-00002. PMID 3342622
- [Background] Ospina-Tascon GA, Bautista DF, Madrinan HJ, Valencia JD, Bermudez WF, Quinones E, Calderon-Tapia LE, Hernandez G, Bruhn A, De Backer D. Microcirculatory dysfunction and dead-space ventilation in early ARDS: a hypothesis-generating observational study. Ann Intensive Care. 2020 Mar 24;10(1):35. doi: 10.1186/s13613-020-00651-1. PMID 32211957